CLINICAL TRIAL: NCT01020149
Title: Evaluation of Nerve Regeneration After Nerve Transsection Using (Diffusion-tensor Magnetic Resonance Imaging) DTI MR Imaging
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Gustav Andreisek, md, University of Zurich
Other Study IDs: 003
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Nerve Degeneration
Keywords: Nerve transsection
MeSH Terms: conditions — Nerve Degeneration | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MR Imaging — MRI is used to evaluate nerve regeneration after traumatic transsection and nerve repair.

SUMMARY:
To prospectively evaluate the nerve regeneration after traumatic nerve transsection using diffusion tensor magnetic resonance imaging (DTI MR imaging).

ELIGIBILITY:
Inclusion criteria:

* Patients with traumatic nerve transsection and nerve repair.

Exclusion criteria:

* contraindication for MRI;
* pregnancy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland